CLINICAL TRIAL: NCT07073404
Title: Omalizumab for the Monotherapy Treatment of Patients With Allergy to Foods of Plant Origin Due to Sensitization to Lipid Transfer Proteins (LTPs) and Profilin
Brief Title: Omalizumab for Plant-Food Allergy Due to Sensitization to LTP or Profilin
Acronym: Omlyclo
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Collaborators: Institute of Biomedical Research in Málaga (IBIMA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Omalizumab proyect
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Food Allergies
Keywords: Omalizumab; FOOD ALLERGIES; LTP; Profilins; Allergy desensitization; Lipid transfer proteins
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be collected at baseline (T0), 2 months (T2), and 4-5 months (T4) after initiation of omalizumab treatment. A total of 60 mL of peripheral blood will be obtained per timepoint: 10 mL in serum separator tubes for humoral studies, 10 mL in lithium heparin tubes for basophil activation test (BAT), and the remaining volume processed using Ficoll gradient for isolation and cryopreservation of peripheral blood mononuclear cells (PBMCs) in liquid nitrogen for future cellular and genomic analyses. Immunological assays include measurement of total and specific IgE and IgG4 to Pru p 3 and Pho d 2 (via ImmunoCAP), and basophil activation test (BAT) analyzed by flow cytometry. Samples may be used for further omics or genetic studies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Omalizumab Injection — Treatment with omalizumab in monotherapy for 16 weeks in patients allergic to vegetables due to sensitization to lipid transfer proteins (LTPs) and profilin.
  Other Names: Omlyclo

SUMMARY:
Omalizumab has demonstrated efficacy, increasing the tolerance threshold in patients with multiple food allergies, as well as reducing the risk of severe reactions when used as monotherapy. This favors improving the reactivity profile of patients with food allergy. In our setting, plant allergy caused by sensitization to panallergens such as lipid transfer proteins (LTPs) and profilins entails important limitations for the consumption of a healthy diet due to the extensive dietary restrictions.

The main objective of this project is to analyze the efficacy of treatment with omalizumab administered every 2-4/weeks, used in monotherapy in patients with plant allergy due to sensitization to profilin and LTPs and those patients in whom sublingual immunotherapy with Pru p 3 (peach LTP), has not been effective, by performing a before-after study we will evaluate the changes in clinical reactivity to LTP (peach) and profilin (melon) and the changes immunological effect after omalizumab intervention. In addition, we will evaluate the changes in reactivity to at least one food other than peach and melon in the different sensitization profiles.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 14-55 years who sign the informed consent (IC) for the study and Biobank sample storage.
* Allergy to plant foods due to sensitisation to LTP, patients allergic to profilin confirmed by a suggestive clinical history, positive skin tests and specific IgE to Pru p 3 (peach LTP) and Pho d 2 (Phoenix dactylifera profilin).
* Positive oral challenge test (OPT) to peach and at least one other food in patients allergic to LTP and positive oral challenge test to melon and at least one other food in patients allergic to profilin.
* Selection of a group of LTP-allergic individuals with therapeutic failure after treatment with ITSL-Pru p 3.

Exclusion Criteria:

* Pregnancy and lactation.
* Immunological diseases; treatment with immunomodulatory and/or blocking drugs.
* Mental illness, which makes it impossible to follow and adhere to treatment (e.g. major depression, psychosis, etc.).
* Severe atopic dermatitis according to SCORAD 5: FEV1<70% (this test will be carried out as a priority in patients with a previous diagnosis of asthma).
* Inflammation in the oral cavity with severe symptoms, as well as with oral surgery in the previous 7 days.
* Immunotherapy with pollens in the previous 2 years.
* Subjects unable to comply with the schedule of visits during the study, as well as due to the consumption of the food under investigation, for example, due to work difficulties.

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with allergy to plant foods due to sensitisation to LTP and profilin
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in tolerated dose of peach or melon during physician-supervised oral food challenge (PPO) in patients with vegetable allergy due to sensitization to lipid transfer proteins (LTPs) or profilin | 16 weeks
  Clinical efficacy will be assessed by measuring the change in the amount (grams) of peach (in LTP-allergic patients) or melon (in profilin-allergic patients) tolerated during a physician-supervised oral food challenge (PPO) after 16 weeks of omalizumab monotherapy. The oral food challenge will be conducted according to standardized EAACI protocols, and the maximum tolerated dose without objective symptoms will be recorded.

SECONDARY OUTCOMES:
To analyze the changes induced in the immunological profile after the intervention: -Humoral: IgE and IgG4 levels to peach LTP (Pru p 3) and palm tree profilin (Pho d 2) by immunoassays. | 16 weeks
To analyze the changes induced in the immunological profile after the intervention: 2.2-Cellular: activation of peach LTP basophils (Pru p 3) and palm profilin (Pho d 2) by flow cytometry. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: María José Torres Jaén, MD, PhD, Principal Investigator — Hospital Regional de Malaga

IPD SHARING:
Plan to Share IPD: Undecided